CLINICAL TRIAL: NCT05727644
Title: Investigation of Pharmacokinetics, Safety and Tolerability of a Single Subcutaneous Dose of NNC0194-0499 in Participants With Various Degrees of Renal Impairment and Normal Renal Function
Brief Title: A Research Study Looking Into Blood and Urine Levels of the Medicine NNC0194-0499 in the Body and How Well it is Tolerated in Participants With Reduced Kidney Function and Normal Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9500-4620; U1111-1277-3646 (Other: World Health Organization (WHO)); 2022-001849-20 (EudraCT Number)
Record Dates: First submitted 2023-02-05; First posted 2023-02-14 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with normal renal function (Active Comparator): Participants will receive a single subcutaneous injection of 30 mg NNC0194-0499.
  Interventions: Drug: NNC0194-0499
- Participants with impaired renal function (Experimental): Participants will receive a single subcutaneous injection of 30 mg NNC0194-0499.
  Interventions: Drug: NNC0194-0499

INTERVENTIONS:
Drug: NNC0194-0499 — Participants will receive a single subcutaneous injection of 30 mg NNC0194-0499.

SUMMARY:
Novo Nordisk is developing the study medicine NNC0194-0499 for the treatment of non-alcoholic steatohepatitis (NASH). NASH is a serious disease where fat, inflammation and scar tissue builds up in the liver. In this study the blood and urine levels of NNC0194-0499 will be compared in people with various degrees of reduced kidney function to the blood and urine levels in people with normal kidney function, after administration of one dose of 30 milligrams (mg) NNC0194-0499. Participant will only get the study medicine in one injection into a skinfold in the thigh (subcutaneous). The study will last for about 66 days including a screening phase of up to 28 days prior to dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-80 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 18.5-39.9 kilogram per meter square (kg/m2) (both inclusive).
* Meeting the pre-defined estimated glomerular filtration rate (eGFR) values based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation according to Kidney Disease: Improving Global Outcomes (KDIGO) 20121, 2 standardized to the individual body surface area (BSA).

Group description eGFR (mL/min)

1. Normal renal function greater than or equal to 90
2. Mild renal impairment 60 - 89
3. Moderate renal impairment 30 - 59
4. Severe renal impairment 15 - 29 not requiring dialysis
5. End-Stage Renal Disease (ESRD) less than 15 or requiring dialysis treatment Renal group 5 (ESRD).

   * Participants requiring dialysis treatment should be on treatment with haemodialysis.

Exclusion Criteria:

* Any disorder, except for conditions associated with renal impairment, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Use of prescription medicinal products or non-prescription drugs, or non-routine vitamins, which at the investigators judgement may affect participant safety or the results of the study within 14 days before screening. Use of the following are allowed: Routine vitamins, occasional use of paracetamol, ibuprofen and topical medication not reaching systemic circulation.
* Use of drugs known to affect creatinine clearance including cephalosporin and aminoglycoside antibiotics, flucytosine, cisplatin, cimetidine, trimethoprim, cibenzoline and nitrofurantoin within 14 days or 5 half-lives, whichever is greater, before planned dosing of the investigational medicinal product (IMP).
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, gastrointestinal, or endocrinological conditions (except conditions associated with renal impairment or ESRD).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
AUC0499,0-∞,SD: Area under the NNC0194-0499 serum concentration-time curve after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of study visit (Visit 9, Day 36)
  Measured as hours*nanomoles per litre (h*nmol/L)

SECONDARY OUTCOMES:
Cmax,0499,SD: Maximum observed serum NNC0194-0499 concentration after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of study visit (Visit 9, Day 36)
  Measured as nanomoles per litre (nmol/L)
tmax,0499,SD: Time to maximum observed serum NNC0194-0499 concentration after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of study visit (Visit 9, Day 36)
  Measured in hours (h)
t½,0499,SD: Terminal half-life of NNC0194-0499 after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of study visit (Visit 9, Day 36)
  Measured in hours (h)
Vz/F0499,SD: Apparent volume of distribution of NNC0194-0499 after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of study visit (Visit 9, Day 36)
  Measured as Litre (L)
CL/F0499,SD: Apparent clearance of NNC0194-0499 after a single dose | From baseline (Visit 2, Day 1, pre-dose) until completion of the end of study visit (Visit 9, Day 36)
  Measured as Litre per hour (L/h)
CLR,0499,SD: Renal clearance of NNC0194-0499 after a single dose | From baseline (Visit 2, Day 1, predose) until completion of the urine collection period 96 hours after dosing (Visit 2, Day 5)
  Measured as Litre per hour (L/h)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com